CLINICAL TRIAL: NCT01884376
Title: Klinische Interventionsstrategie Zur überbrückenden Behandlung Peripherer Nervendefekte Mit Neuromaix
Brief Title: Clinical Study for the Treatment of Peripheral Nerve Defects With Neuromaix
Acronym: PeRepair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-009
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Patients With a Scheduled (Diagnostic) Nervus Suralis Biopsy
Keywords: nerve biopsy; nerve regeneration; neuroma pain; loss of sensation
MeSH Terms: conditions — Disease; Hypesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neuromaix implantation (Experimental): Implantation of Neuromaix during an diagnostic nerve biopsy
  Interventions: Device: Neuromaix

INTERVENTIONS:
Device: Neuromaix

SUMMARY:
The aim of this study is the development and initial clinical application of the nerve guide Neuromaix in humans to provide evidence for the safety and performance of the device.

Neuromaix is intended to be used as a guiding structure to bridge a peripheral nerve discontinuity, and to create a conduit for axonal growth across the nerve gap.

DETAILED DESCRIPTION:
The Neuromaix nerve guide is an absorbable implant composed of porcine collagen, used to bridge a peripheral nerve discontinuity, and to create a conduit for axonal growth across the nerve gap. Neuromaix provides a protective environment for peripheral nerve regeneration after injury. Neuromaix connects the proximal and distal ends of a transected nerve, allowing regenerating axons to grow through the scaffold, into the distal nerve tissue towards the target muscle or skin.

Neuromaix is composed of two parts. The Epimaix part provides the structural characteristics needed to suture the nerve guide in place and to prevent ingrowth of scar tissue. The Perimaix part provides a structure that mimics endoneurial tubes, providing guidance for the regenerating axons while bridging the nerve gap.

ELIGIBILITY:
Inclusion Criteria:

* both genders in the age between 18 und 70 years
* patients who are scheduled for a nerve biopsy

Exclusion Criteria:

* alcohol-related polyneuropathy
* paraneoplastic polyneuropathy
* present: immunosuppressive therapy
* present: malignant tumor
* peripheral vascular diseases
* collagen diseases (e.g. existing keloid scars)
* patients with an increased wound healing disorder (e.g. diabetics)
* patients with chronic venous insufficiency (vein thrombosis, skin diseases)
* patients with coagulation and bleeding disorders (ASA- or Marcumar-patients)
* present: pregnancy
* HIV, Hepatitis B or Hepatitis C infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
proof of safety of the medical device Neuromaix | 12 months
  The primary objective is the proof of safety of the medical device Neuromaix. key parameter: normal wound healing without complications

SECONDARY OUTCOMES:
effectiveness evaluation of the implant device Neuromaix | 12 months
  The secondary objective is the evaluation of the effectiveness of the Neuromaix implantation ("Performance arm of study").
  key parameters: axonal regeneration and recovery of sensory function

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Bozkurt, PD Dr. med., Principal Investigator — Department of Plastic Surgery, Hand Surgery and Burn Center,University Hospital RWTH Aachen
Locations (1):
- Department of Plastic Surgery, Hand Surgery and Burn Center, University Hospital RWTH Aachen, Aachen, Germany